CLINICAL TRIAL: NCT07352995
Title: Colonoscopic Investigation of the Correlation Between Bowel Wall Inflammation and Luminal Temperature Rise in IBD
Brief Title: Thermal Measurements of the Gut With a Colonoscope Compatible Thermal Probe
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Principal Investigator, Guillermo Tearney, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2025P000709
Record Dates: First submitted 2026-01-13; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- IBD, Crohn's Disease, and/or UC (Experimental): 10 adult participants currently diagnosed with inflammatory bowel disease (IBD), Crohn's disease, and/or ulcerative colitis (UC) will be enrolled at MGH
  Interventions: Device: Feasibility of using a thermal probe to measure temperature rise in colonic mucosa
- Undergoing Colorectal Screening (Experimental): 10 adult subjects undergoing colorectal cancer screening will be enrolled at MGH
  Interventions: Device: Feasibility of using a thermal probe to measure temperature rise in colonic mucosa

INTERVENTIONS:
Device: Feasibility of using a thermal probe to measure temperature rise in colonic mucosa — 10 participants in each arm will be enrolled in this study. All consented participants will receive the same intervention.

SUMMARY:
The goal of this clinical trial is to use a modified thermal probe to measure temperature rise in the colonic mucosa of participants with inflammatory bowel disease, Crohn's disease, and/or ulcerative colitis. The main question it aims to answer is:

Is the thermal probe an effective device to use to detect temperature rise in the colonic mucosa?

During the participant's standard of care colonoscopy, the thermal probe will be inserted into the colonoscope. The thermal probe is connected to a temperature transmitter that collects and saves the temperature of the colon in real time.

ELIGIBILITY:
Inclusion Criteria:

* Participants 18 years or older
* Participants undergoing elective colonoscopy
* Participants capable of following requirements
* Participants capable of providing informed consent
* Participants with a diagnosis of IBD, Crohn's disease, and/or ulcerative colitis or participants undergoing colorectal cancer screening

Exclusion Criteria:

* Participants contraindicated for colonoscopy, including experiencing acute events within the last 6 weeks prior to the colonoscopy (i.e. subjects suffering from a myocardial infarction (heart attack), diagnosis of peritonitis (the inflammation of the membrane lining of the abdominal wall), diagnosis of hemodynamic instability (shock), surgery involving colonic anastomosis (reconnection of the colon), and/or bowel injury (from trauma or surgery)
* Participants who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Ability of thermal probe to collect temperature measurements from colonic mucosa | Thermal measurements are collected during the study procedure and analyzed within one year of collection.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Tearney, M.D., PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States